CLINICAL TRIAL: NCT01401933
Title: A Phase 1 Study To Assess the Effect of Rifampin on the Pharmacokinetics of Linifanib in Subjects With Advanced or Metastatic Solid Tumors
Brief Title: Effect of Rifampin on the Pharmacokinetics of Linifanib in Subjects With Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: M11-307
Record Dates: First submitted 2011-04-29; First posted 2011-07-26 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-10

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — linifanib; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Linifanib (Experimental)
  Interventions: Drug: Linifanib; Drug: Rifampin

INTERVENTIONS:
Drug: Linifanib — QD on Days 1 and 13
  Other Names: ABT-869
Drug: Rifampin — QD on Days 5-16
  Other Names: Rifadin

SUMMARY:
This is a phase 1, open-label study designed to determine the interaction of rifampin with linifanib.

DETAILED DESCRIPTION:
This study is designed to explore the drug interaction between rifampin and linifanib to determine the potential effect of rifampin on the metabolism of linifanib. Linifanib will be taken alone or in combination with rifampin. The safety of a single dose administration of linifanib when administered alone and in combination with rifampin will be assessed. Subjects may enroll in a separate extension study to continue receiving linifanib after completion of this study.

ELIGIBILITY:
Inclusion Criteria

1. Age is greater than or equal to 18 years.
2. Subject must have a histologically or cytologically confirmed non-hematologic malignancy other than HCC.
3. Eastern Cooperative Oncology Group (ECOG) Performance Score of 0-2.
4. Subject must have adequate bone marrow, renal and hepatic function.

   * Bone Marrow: Absolute neutrophil count (ANC) >= 1,500/mm^3 (1.5 X 10^9/L); Platelets >= 75,000/mm^3 (75 X 10^9/L); Hemoglobin >= 9.0 g/dL (1.4 mmol/L)
   * Renal function: serum creatinine <= 2.0 mg/dL (0.81 mmol/L);
   * Hepatic function: AST and ALT <= 1.5 X ULN unless liver metastases are present, then AST and ALT <= 5.0 X ULN; bilirubin <= 1.5 mg/dL (0.026 mmol/L).
5. Subject must have Partial Thromboplastin Time (PTT) </= 1.5 X Upper Limit of Normal ( ULN) and International Normalized Ratio (INR) </= 1.5.

Exclusion Criteria

1. Subject has received anti-cancer therapy including investigational agents, cytotoxic chemotherapy, radiation therapy or biologic therapy within 21 days or within a period defined by 5 half lives, whichever is shorter, prior to study drug administration. In addition subject has not recovered to less than or equal to Grade 1 clinically significant adverse effects/toxicities of the previous therapy.
2. Subject has undergone major surgery within 21 days of Study Day 1.
3. Subject has untreated brain or meningeal metastases. Subjects with treated brain metastases that are radiographically or clinically stable (for at least 4 weeks after therapy) and who have no evidence of cavitation or hemorrhage in the brain lesion, are eligible provided that they are asymptomatic and do not require corticosteroids (must have discontinued steroids at least 1 week prior to Study Day 1).
4. Subject has received potential inhibitors of the metabolism of linifanib within 21 days prior to initial study drug administration. Such drugs include CYP3A inhibitors, CYP1A2 inhibitors, CYP2C19 inhibitors, CYP2C8 substrates and CYP3A inducers.
5. Current enrollment in another clinical trial..

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To investigate the effect of rifampin on the pharmacokinetic of linifanib in subjects with advanced or metastatic solid tumors. | Blood samples for the PK of linifanib will be collected at various time points from Day 1 through Day 17.
  To assess the effect of rifampin on the pharmacokinetics of linifanib and metabolite(s), an analysis will be performed for the natural logarithms of Cmax and AUC of linifanib and metabolite(s) with concentrations that permit confident determination of values of the pharmacokinetic variables. A paired t-test will be performed to compare the central value on Study Day 13 (with rifampin) to that on Study Day 1 (without rifampin). Point estimates and 90% confidence intervals will also be provided.

SECONDARY OUTCOMES:
Safety: Adverse Events - The number of participants with adverse events will be reported as a measure of Safety. | Through out the study
  The investigators will monitor each subject for clinical and lab evidence of adverse events on a routine basis through out the study.
Safety: Physical Examination and Vital Signs - Physical examination will be performed and vital signs will be assessed for participants as a measure of safety. | Physical exam will be done at Screening, Day1, Day 13, Day 17/Final Visit and 30 day safety follow-up. Vital Signs (blood pressure, heart rate, body temperature) will be done at all visits.
  Complete physical exam, including body weight, will be done at Screening and Day 1. A symptom-directed physical exam, including weight, will be done at Day 13, Day 17/Final Visit and 30 day safety follow-up.
Safety: Clinical Lab Tests will be performed for each participant as a safety measure. | Screening, Day 1, Day 13, Day 17/Final Visit and 30 day safety follow up visit.
  Chemistry, hematology, urinalysis lab tests.

CONTACTS AND LOCATIONS:
Overall Officials: Mark D. McKee, MD, Study Director — Abbott
Locations (2):
- United States (2):
  - Site Reference ID/Investigator# 49953, Tucson, Arizona
  - Site Reference ID/Investigator# 49952, Madison, Wisconsin